CLINICAL TRIAL: NCT02698501
Title: Effects of Anti-TSLP on Airway Hyperresponsiveness and Mast Cell Phenotype in Asthma - A Randomized Double-blind, Placebo-controlled Trial of MEDI9929
Brief Title: Effects of Anti-TSLP in Patients With Asthma
Acronym: UPSTREAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celeste Porsbjerg (Other)
Collaborators: Lund University (Other); University of Newcastle, Australia (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Celeste Porsbjerg, Chief Physician, PhD, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-15-10870
Record Dates: First submitted 2016-02-05; First posted 2016-03-03 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Asthma
Keywords: Asthma; Airway hyperresponsiveness; TSLP; Mast cell; Eosinophil
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI9929 (Experimental): MEDI9929 is a human monoclonal antibody immunoglobulin IgG2λ directed against TSLP. MEDI9929 binds with human TSLP and prevents its interaction with thymic stromal lymphopoietin receptor (TSLPR).
  Interventions: Drug: MEDI9929
- Placebo (Placebo Comparator): Apart from the active substance, the placebo is otherwise identical to IMP.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI9929 — MEDI9929 700mg (3 doses in total, 4-week intervals), administered intravenously
  Arms: MEDI9929
Drug: Placebo — Placebo (3 doses in total, 4-week intervals), administered intravenously
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether anti-TSLP will decrease airway hyperresponsiveness in patients with asthma already on daily treatment with inhaled corticosteroids.

The investigators expect that airway hyperresponsiveness will decrease after treatment with anti-TSLP, and that this happens due to a change in the type of mast cells with in the lungs. Also, the investigators expect a decrease in inflammatory cells and mediators measured in material from the lungs.

Half of the participants will receive anti-TSLP (MEDI9929) on top of their regular asthma treatment, while the other half will receive placebo on top of their regular asthma treatment.

DETAILED DESCRIPTION:
The mannitol test is increasingly used by clinicians to diagnose asthma. It has clinical advantages in terms of being feasible in a wide range of settings with the need of a minimum of equipment. Airway hyper responsiveness (AHR) to mannitol correlates with eosinophilic airway inflammation and the degree of asthma control, predicts the risk of exacerbation and response to inhaled steroids.

Subjects with asthma and indirect AHR have increased levels of intraepithelial carboxypeptidase A3 (CPA3), a metalloexopeptidase specifically expressed by mast cells, compared to asthmatics without AHR. CPA3 is known to be selectively present in the MCTC phenotype (mast cells containing both tryptase and chymase), and recent studies suggest that increased CPA3 levels also constitutes a marker of a Th2-high/eosinophilic and steroid-responsive asthma. Interestingly, treating mast cell precursors with TSLP increases CPA3 immunostaining, suggesting that TSLP released by e.g. airway epithelium up-regulate a mast cell phenotype that is potentially important in AHR and also promotes eosinophilic airway inflammation. Previous published data by the investigators confirm that increased MCTC in submucosa of subjects with asthma is associated with an increased CPA3 and TSLP expression.

The investigators speculate that the effect of MEDI9929 on AHR to mannitol is likely to be primarily a consequence of functional differences in mast cells. Treating subjects with asthma with MEDI9929 will potentially block downstream effects on mast cell activation as well as eosinophilic inflammation, which may reduce AHR to inhaled mannitol.

The purpose of this study is to investigate whether AHR to mannitol is a suitable marker of response to MEDI9929, but also to better understand the anti-inflammatory effects of MEDI9929 in the lungs, including whether a reduced AHR to mannitol following treatment with MEDI9929 is related to a reduction in chymase/CPA-3 positive mast cells. The investigators hypothesize that MEDI9929 will decrease the response to mannitol (measured as an increase in PD15) after 12 weeks of treatment as compared to placebo. It is further hypothesized that the number of chymase/CPA-3 positive mast cells in airway epithelium and submucosa will be reduced after 12 weeks of treatment with MEDI9929 in subjects with AHR to mannitol.

This trial offers the opportunity to study potential biomarkers and surrogate endpoints, but also to identify the anti-inflammatory effects of MEDI9929 on a mechanistic level.

This study is a randomized, double-blind, placebo-controlled trial. It includes a enrolment period of maximum 2 weeks, 12 weeks of treatment (three IV doses of either 700mg MEDI9929 or placebo) and 8 weeks follow-up after the second bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age 18 through 75, inclusive at the time of Visit 1
3. Body mass index between 18-40 kg/m2 (both inclusive) and weight ≥ 40 kg at Visit 1.
4. A diagnosis of asthma as defined by GINA (ginasthma.org).
5. ICS (in any dose) on a daily basis for at least three months prior to Visit 1
6. A stable asthma controller regimen with ICS (±LABA) for at least 4 weeks prior to Visit 1
7. A FEV1 value of ≥ 70% at Visit 1
8. ACQ-6 > 1 (partly controlled) at Visit 1
9. PD15 to mannitol <= 315 mg at visit 1
10. Subjects must demonstrate acceptable inhaler and spirometry techniques during screening (as evaluated and in the opinion of study site staff)
11. Subjects must demonstrate ≥ 70% compliance with usual asthma controller ICS±LABA during the screening (V1 to V3).

Exclusion Criteria:

1. Current smokers or subjects with a smoking history of ≥ 10 pack years. Former smokers with < 10 pack years must have stopped for at least 6 months to be eligible.
2. Previous medical history or evidence of an uncontrolled intercurrent illness.
3. Any concomitant respiratory disease that in the opinion of the investigator and/or medical monitor will interfere with the evaluation of the investigational product or interpretation of subject safety or study results.
4. Clinically relevant abnormal findings in hematology or clinical chemistry.
5. Evidence of active liver disease.
6. History of cancer.
7. Acute upper or lower respiratory infections.
8. Helminth parasitic infection.
9. Known history of active tuberculosis (TB).
10. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology.
11. A positive human immunodeficiency virus (HIV) test.
12. History of sensitivity to any component of the investigational product.
13. History of anaphylaxis to any biologic therapy.
14. History of documented immune complex disease (Type III hypersensitivity reactions) to mAb administration.
15. History of any known primary immunodeficiency disorder.
16. Oral corticosteroids.
17. Use of 5-lipoxygenase inhibitors.
18. Use of immunosuppressive medication.
19. Pregnant, breastfeeding or lactating females.
20. History of chronic alcohol or drug abuse.
21. Receipt of the Th2 cytokine inhibitor suplatast
22. Receipt of any live or attenuated vaccines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Decrease in airway hyperresponsiveness to mannitol in response to treatment with MEDI9929 in patients with asthma | 12 weeks
  Change in PD15 to mannitol (provoking dose for 15% reduction in FEV1, expressed as doubling doses) measured at baseline and after the 12-week treatment period between groups.
Supportive primary objective 1: Mannitol test negative in response to treatment with MEDI9929 in patients with asthma | 12 weeks
  Number of mannitol test negative (PD15 > 635mg) subjects after a 12-week treatment period between groups
Supportive primary objective 2: Decrease in airway hyperresponsiveness to mannitol in response to treatment with MEDI9929 in patients with asthma | 12 weeks
  The change in PD15 to mannitol measured at baseline and after the 12-week treatment period, expressed as geometric mean calculated by linear interpolation, compared between treatments.
Supportive primary objective 3: Decrease in airway hyperresponsiveness to mannitol in response to treatment with MEDI9929 in patients with asthma | 12 weeks
  Change in RDR (Response Dose Ratio) to mannitol measured at baseline and after the 12-week treatment period between groups

SECONDARY OUTCOMES:
Change in number of Chymase/CPA-3 positive mast cells following treatment with MEDI9929 | 12 weeks
  Cell count (MCT, MCTC and MCCPA3) in airway submucosa, airway epithelium and airway smooth muscle measured at baseline and after the 12-week treatment period between groups
Changes in percentage of airway eosinophils and neutrophils in sputum in patients treated with MEDI9929 compared to placebo. | 12 weeks
  Percentage of eosinophils and neutrophils in sputum measured at baseline and after the 12-week treatment period.
Changes in percentage of airway eosinophils and neutrophils in airway submucosa in patients treated with MEDI9929 compared to placebo. | 12 weeks
  Percentage of eosinophils and neutrophils in airway submucosa measured at baseline and after the 12-week treatment period.
Changes in number of airway eosinophils and neutrophils in blood in patients treated with MEDI9929 compared to placebo. | 12 weeks
  Number of eosinophils and neutrophils in blood, measured at baseline and after the 12-week treatment period.

OTHER OUTCOMES:
Change in diversity in airway microbiota in patients treated with MEDI9929 compared to placebo | 12 weeks
  Diversity of airway microbiota as measured by 16S gene sequencing in BAL measured at baseline and after the 12-week treatment period
Change in airway microbiota in patients treated with MEDI9929 compared to placebo | 12 weeks
  Relative abundances of airway microbiota as measured by 16S gene sequencing in BAL measured at baseline and after the 12-week treatment period
The effect of MEDI9929 on TSLP mRNA expression | 12 weeks
  mRNA expression of TSLP in airway submucosa, airway epithelium and sputum.
The effect of MEDI9929 on IL-33 mRNA expression | 12 weeks
  mRNA expression of IL-33 in airway submucosa, airway epithelium and sputum.
The effect of MEDI9929 on TLRs mRNA expression | 12 weeks
  mRNA expression of TLRs in airway submucosa, airway epithelium and sputum.
The effect of MEDI9929 on IL-4 mRNA expression | 12 weeks
  mRNA expression of IL-4 in airway submucosa, airway epithelium and sputum.
The effect of MEDI9929 on IL-5 mRNA expression | 12 weeks
  mRNA expression of IL-5 in airway submucosa, airway epithelium and sputum.
The effect of MEDI9929 on IL-13 mRNA expression | 12 weeks
  mRNA expression of IL-13 in airway submucosa, airway epithelium and sputum.
The effect of MEDI9929 on level of Fractional Exhaled Nitric Oxide (FeNO) | 12 weeks
  Level of FeNO (ppb) before and after 12-weeks treatment between groups
The effect of MEDI9929 on use of rescue medication | 12 weeks
  Number of puffs / week measured at baseline and after the 12-week treatment period
Frequency of ILC2s in peripheral blood before and after treatment | 12 weeks
  Number of ILC2 in peripheral blood measured at baseline and after the 12-week treatment period between groups
Adverse Events | up to 28 weeks
  number of reported Adverse Events between groups
Change in ACQ | 12 weeks
  ACQ-score measured at baseline and after the 12-week treatment period between groups
Change in lung function | 12 weeks
  FEV1 (post beta2) measured at baseline and after the 12-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Porsbjerg, MD, PhD, Principal Investigator — Copehagen University Hospital Bispebjerg, Copenhagen, Denmark
Locations (1):
- Copenhagen University Hospital Bispebjerg, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sverrild A, Hansen S, Hvidtfeldt M, Clausson CM, Cozzolino O, Cerps S, Uller L, Backer V, Erjefalt J, Porsbjerg C. The effect of tezepelumab on airway hyperresponsiveness to mannitol in asthma (UPSTREAM). Eur Respir J. 2021 Dec 31;59(1):2101296. doi: 10.1183/13993003.01296-2021. Print 2022 Jan. No abstract available. PMID 34049943